CLINICAL TRIAL: NCT07392294
Title: Comparison of Foam Dressing Versus Silver-Impregnated Foam Dressing for Prevention of Peristomal Complications in Pediatric Tracheostomy: A Prospective Randomized Controlled Trial Using Validated Assessment Tools
Brief Title: Foam Dressing Versus Silver Foam Dressing for Pediatric Tracheostomy Wound Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem Atasehir Hospital (Other)
Responsible Party: Principal Investigator, SERAP SAHIN ONDER, associate professor, Acibadem Atasehir Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 85-2021; 2022/001). (Other Grant/Funding Number: Science Research Program of Health Sciences University.)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Tracheostomy Complication; Pressure Ulcer (PU); Surgical Wound
Keywords: Pediatric tracheostomy; Foam dressing; Silver-impregnated dressing; Pressure ulcer prevention; Peristomal complications; Wound care; Braden Q Scale; Children
MeSH Terms: conditions — Pressure Ulcer; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Foam Dressing (Active Comparator): Patients received standard foam dressing for tracheostomy wound care (Group A, n=25)
  Interventions: Device: Standard Foam Dressing
- Silver-Impregnated Foam Dressing (Experimental): Patients received silver-impregnated foam dressing for tracheostomy wound care (Group B, n=25)
  Interventions: Device: Silver-Impregnated Foam Dressing

INTERVENTIONS:
Device: Standard Foam Dressing — DescriptionStandard foam dressing applied under tracheostomy cannula. Dressings were changed when 75% saturated with secretions or left in place up to 7 days if dry.
  Arms: Standard Foam Dressing
Device: Silver-Impregnated Foam Dressing — Silver-impregnated foam dressing applied under tracheostomy cannula. Dressings were changed when 75% saturated with secretions or left in place up to 7 days if dry.
  Arms: Silver-Impregnated Foam Dressing

SUMMARY:
This study compares two types of wound dressings used after tracheostomy surgery in children: standard foam dressing and silver-impregnated foam dressing.

Tracheostomy is a surgical procedure that creates an opening in the neck to help children breathe. Skin problems around the tracheostomy site are common, occurring in up to 29% of pediatric patients.

The purpose of this study is to determine if silver-impregnated foam dressing is better than standard foam dressing in preventing skin complications around the tracheostomy site.

Fifty children (ages 0-18 years) undergoing tracheostomy surgery were randomly assigned to receive either standard foam dressing or silver-impregnated foam dressing. All patients received the same standardized wound care. Patients were followed for one month after surgery.

The main outcome measured was the rate of skin complications. Secondary outcomes included pressure ulcer risk assessment using the Braden Q Scale and wound staging using the National Pressure Injury Advisory Panel classification.

DETAILED DESCRIPTION:
Peristomal skin complications represent a significant concern following pediatric tracheostomy, with reported incidence rates up to 29%. These complications include pressure ulcers, infections, granulation tissue, and skin breakdown.

This prospective randomized controlled trial was conducted at a single tertiary care center. Fifty pediatric patients undergoing elective tracheostomy were enrolled and randomly assigned to one of two groups:

Group A (n=25): Standard foam dressing Group B (n=25): Silver-impregnated foam dressing

All patients received a standardized postoperative care protocol including:

* Velcro ties with foam padding for tube securement
* Daily wound assessment
* Neutral head positioning for ventilated patients
* Standardized dressing change criteria

Patients were assessed on postoperative days 1, 7, 14, 21, and 30. Pressure ulcer risk was evaluated using the Braden Q Risk Assessment Scale, and any pressure injuries were staged according to the National Pressure Injury Advisory Panel (NPIAP) classification system.

This is the first randomized controlled trial comparing these dressing types using validated, standardized assessment tools in pediatric tracheostomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0-18 years
* Undergoing elective tracheostomy
* Tracheostomy performed by the pediatric otolaryngology team
* Followed in neonatal or pediatric intensive care units

Exclusion Criteria:

* Patients over 18 years of age
* Emergency tracheostomy
* Percutaneous tracheostomy
* Pre-existing skin diseases
* History of head and neck surgery
* Tracheostomy performed during airway reconstruction surgery

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Peristomal Complications | 30 days postoperatively
  Measure DescriptionOverall rate of peristomal complications including infection, pressure ulcer, granulation tissue, and skin necrosis. Measured as percentage of patients developing any complication.

SECONDARY OUTCOMES:
Braden Q Risk Assessment Scale Score | Postoperative days 1, 7, 14, and 21
  Measure DescriptionPressure ulcer risk assessment using Braden Q Scale (score range 7-28). Lower scores indicate higher risk: ≤12 high risk, 13-15 moderate risk, ≥16 no risk.
Pressure Ulcer Severity by NPIAP Classification | 30 days postoperatively
  Measure DescriptionPressure ulcer staging according to National Pressure Injury Advisory Panel (NPIAP) classification system: Stage 1 (non-blanchable erythema), Stage 2 (partial-thickness skin loss), Stage 3 (full-thickness skin loss), Stage 4 (full-thickness tissue loss).

CONTACTS AND LOCATIONS:
Overall Officials: Asli SAHIN YILMAZ, professor, Study Chair — Umraniye Education and Research Hospital
Locations (1):
- Acibadem Atasehir Hastanesi, Istanbul, Ataturk Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.